CLINICAL TRIAL: NCT01861067
Title: A Randomized Comparison of Laparoendoscopic Single-site (LESS) Hysterectomies: Total Laparoscopic Hysterectomy (TLH) Versus Laparoscopically Assisted Vaginal Hysterectomy (LAVH)
Brief Title: LESS-TLH Versus LESS-LAVH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KNC13-014
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Benign Uterine Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LESS-TLH (Experimental): laparoendoscopic single-site (LESS) total laparoscopic hysterectomy (TLH)
  Interventions: Procedure: LESS-TLH
- LESS-LAVH (Active Comparator): laparoendoscopic single-site (LESS) laparoscopically-assisted vaginal hysterectomy (LAVH)
  Interventions: Procedure: LESS-LAVH

INTERVENTIONS:
Procedure: LESS-TLH
  Arms: LESS-TLH
Procedure: LESS-LAVH
  Arms: LESS-LAVH

SUMMARY:
During the last 2 decades, several studies have tried to define the best surgical approach to hysterectomy for benign uterine diseases1. Accumulating evidence demonstrates that abdominal hysterectomy has a higher incidence of complications, a longer hospital stay and a slower convalescence in comparison with laparoscopic hysterectomy (LH). The main advantage of LHs is the absence of a wide abdominal scar, which results in fewer wound-related complications and in a significant decrease of postoperative pain.

Technologic advances in endoscopic instrumentation and optics have allowed the development of an even less invasive procedure than conventional LH using multiple ports: laparoendoscopic single-site (LESS) surgery, also known as single-port access (SPA) laparoscopy3. In the LESS approaches, total laparoscopic hysterectomy (TLH) and laparoscopically-assisted vaginal hysterectomy (LAVH) are all feasible, with comparable conventional LH. However, it is yet to be determined which of two alternative and less invasive approaches (LESS-TLH and LESS-LAVH) should be preferred. In particular, none has focused on postoperative pain as the primary outcome of the study. The investigators have therefore designed the randomized trial to investigate specifically differences in postoperative pain after LESS-TLH and LESS-LAVH.

ELIGIBILITY:
Inclusion Criteria:

* women with indication for hysterectomy for a supposed benign uterine disease
* women with an age of 18 years or older
* women who were not pregnant at the time of presentation
* women who were appropriated medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification 1 or 2)

Exclusion Criteria:

* uterine volume > 18 weeks of gestation by pelvic examination
* suspicion of malignancy
* pelvic organ prolapse > stage 1 according to POP-Q classification
* inability to understand and provide written informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Operative time | Surgery date
  Operative time was defined as the time from skin incision to skin closure, which was electronically recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — CHA Gangnam Medical center
Locations (1):
- CHA Gangnam Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song T, Kim MK, Kim ML, Jung YW, Yun BS, Seong SJ. A Randomized Comparison of Laparoendoscopic Single-Site Hysterectomies: Total Laparoscopic Hysterectomy Versus Laparoscopically Assisted Vaginal Hysterectomy. J Laparoendosc Adv Surg Tech A. 2015 Jul;25(7):541-7. doi: 10.1089/lap.2014.0524. Epub 2015 Jun 15. PMID 26075931